CLINICAL TRIAL: NCT06839469
Title: Establishing Walking-related Digital Biomarkers in Rare Childhood Onset Progressive Neuromuscular Disorders
Status: Recruiting | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: Stevens Institute of Technology (Other); Stanford University (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Boston Children's Hospital, Boston, MA, USA (Other)
Responsible Party: Principal Investigator, Jacqueline Montes, Principal Investigator, Columbia University
Other Study IDs: AAAU9807; R01HD112908 (NIH)
Record Dates: First submitted 2025-02-17; First posted 2025-02-21 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-02

CONDITIONS: Spinal Muscular Atrophy Type 3; Duchenne Muscular Dystrophy (DMD)
Keywords: SMA; spinal muscular atrophy; duchenne muscular dystrophy; DMD; instrumented insole; neuromuscular disease; machine learning model; gait analysis; functional biomarker; wearable; six minute walk test; ambulatory; becker phenotype
MeSH Terms: conditions — Spinal Muscular Atrophies of Childhood; Muscular Dystrophy, Duchenne; Muscular Atrophy, Spinal; Neuromuscular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Spinal Muscular Atrophy: Ambulatory children and adults at least 5 years old by the time of enrollment with genetically confirmed SMA.
- Duchenne Muscular Dystrophy: Ambulatory children and adults ages at least 5 years old by the time of enrollment with genetically confirmed Duchenne or Becker muscular dystrophy or evidence on muscle biopsy with a clinical presentation consistent with DMD/BMD.
- Healthy Control: The healthy control group will be ambulatory children and adults at least 5 years of age, age- and gender-matched to the SMA and DMD groups as best as possible.

SUMMARY:
The purpose of this research is (1) to identify disease specific walking-related digital biomarkers of disease severity, and (2) monitor longitudinal changes in natural environments, for extended periods of time, in DMD and SMA.

DETAILED DESCRIPTION:
Spinal muscular atrophy (SMA) and Duchenne muscular dystrophy (DMD) are genetic disorders that often result in progressive weakness and impaired function. Our recent findings suggest that novel machine-learning (ML)-based abstraction models may map noisy signals from foot-worn sensors (namely, instrumented insoles developed by the project team) into accurate and clinically relevant spatiotemporal and kinetic gait parameters. These gait parameters derived from instrumented insoles may serve as functional biomarkers to detect changes in real world function. All participants will be observed and measured while wearing the instrumented insoles in the lab and in real-life environments.

ELIGIBILITY:
Inclusion Criteria:

* Genetic confirmation of disease (DMD, SMA) or healthy control
* Able to walk independently at least 25 meters
* Ongoing corticosteroids therapy or initiation of corticosteroid therapy in the previous 3 months for DMD
* Stable dose of FDA approved SMN up-regulator therapy or in an open-label extension phase of a study treatment for at least 6 months for SMA or gene replacement at enrollment for SMA or DMD participants.

Exclusion Criteria:

* Use foot orthoses or assistive devices for community ambulation or a mobility device for community navigation
* Use investigational medications intended for treatment of NMD within 30 days
* Prior to study entry had an injury or surgery that would impact gait within the previous 3 months

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study sample will include 33 ambulatory SMA participants, 33 ambulatory DMD participants, and 40 healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 106 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Six Minute Walk Test | One day
  Participants will complete the six minute walk test in a corridor which includes the instrumented walkway, while wearing the insoles. This is to measure spatial parameters, kinetic parameters, temporal parameters, and metrics of cumulative activity in order to compare against the gold standard instrumented walkway. The six minute walk test is an objective evaluation of functional exercise capacity, and measures the maximum distance a person can walk in six minutes over a 25 meter course.
10 Meter Walk/Run | One day
  Participants will walk, or run if able to, for 10 meters on the instrumented walkway while also wearing the insoles. This will be done to measure spatial parameters, kinetic parameters, temporal parameters, and metrics of cumulative activity in order to compare against the gold standard instrumented walkway. This outcome is reported as the time it takes for the participant to complete 10 meters as fast as possible.
Time Up and Go Test (TUG) | One day
  Participants will complete the TUG test. This is a timed test of mobility, requiring the participant to stand up from a seated position, walk 3 meters and return to sitting in the chair. The outcome reported is the time it takes for the participant to complete the sequence.
Muscle Strength Testing with Hand-held Dynamometry (HHD) | One day
  HHD is used to assess the strength of muscles and is reported as the maximum strength exerted in pounds (lbs).
30 Second Sit to Stand Test (30STS) | One day
  30STS test is used to basic muscle power and function. The participant begins seated with their arms at their sides, feet flat on the floor and back against the chair. They are instructed to rise up to a full standing position and sit back down as many times as possible in 30 seconds, with or without using their hands for support.
Ankle Range of Motion | One day
  Ankle range of motion (ROM) will be assessed on both the left right side using standardized goniometers. The procedures used will be standardized and performed by trained physical therapists who have attended in-person training. ROM will be recorded in degrees for plantar flexion and dorsiflexion.
Knee Extension Range of Motion | One day
  Knee extension range of motion (ROM) will be assessed on both the left right side using standardized goniometers. The procedures used will be standardized and performed by trained physical therapists who have attended in-person training. ROM will be recorded in degrees of knee extension.
Hip Extension Range of Motion | One day
  Hip extension range of motion (ROM) will be assessed on both the left right side using standardized goniometers. The procedures used will be standardized and performed by trained physical therapists who have attended in-person training. ROM will be recorded in degrees of hip extension.

SECONDARY OUTCOMES:
Free-living Testing of Instrumented Insoles | One month
  To determine spatial parameters, kinetic parameters, temporal parameters, and metrics of cumulative activity using instrumented insoles, participants with SMA, DMD, and healthy controls will be asked to wear the insoles along with a validated activity tracker. Participants will be asked to wear the insoles during a single day visit to the lab, and then for at least 180 hours at home in a real-life environment. Participants will be asked to wear the insoles and activity tracker for at least 6 hours per day when at home. Compliance with this outcome will be measured in total hours the insoles are worn over the study period (one month).
Validation of Physical Activity using Actigraph accelerometer | One month
  An Actigraph will be provided and worn during waking hours, while the participant is also wearing the insoles. Data extracted are counts per minutes, and are measurements of movement performed in both vertical and horizontal axis. The counts will be used to quantify the time the participant is inactive, low, moderate and / or in vigorous physical active.
International Physical Activity Questionnaire-Short Form, IPAQ-SF | One day
  The IPAQ-SF is a self report questionnaire that assesses the types of intensity of physical activity and sitting time that people do as part of their daily lives. It is used estimate total physical activity in MET-min/week and time spent sitting in the 7 days prior to completing the questionnaire. It will be completed by participants aged 18 and over, at the start and at the end of the one-month insole wear time.
PROMIS Pediatric Physical Activity Questionnaire | One day
  The pediatric activity questionnaire measures a child's self-report of short bouts of moderate to vigorous physical activity. This questionnaire is designed to measure constructs best recalled by children such as physiological response, symptoms, and short bouts of higher intensity activity. The questionnaire has an 8-item bank and is intended for use with children ages 8 to 17 years or with a parent proxy version for children aged 5 to 17 years. It will be completed at the start and at the end of the one month insole wear time and scores will calculated and range from 8-40.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Stanford University, Palo Alto, California
  - Boston Children's Hospital, Boston, Massachusetts
  - Columbia University Irving Medical Center, New York, New York

IPD SHARING:
Plan to Share IPD: Undecided